CLINICAL TRIAL: NCT00712010
Title: Acute Metabolic Effect of the Protein Quality of a High-protein Meal Replacement in Healthy Men
Brief Title: Metabolic Effect of High-protein Meals in Men
Acronym: OPTI-PROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, CDUadmin, Principal Investigator, Société des Produits Nestlé (SPN)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 07.26.MET; Ethics: 71/08
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Results first posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Glucose; Insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Whey protein native (Experimental): Whey protein native versus the 6 other arms
  Interventions: Other: Whey protein microgels; Other: Hydrolyzed whey protein; Other: Casein native; Other: Hydrolyzed casein; Other: Total milk protein native; Other: Hydrolyzed milk protein
- Whey protein microgels (Experimental): Whey protein microgels versus the 6 other arms
  Interventions: Other: Whey protein native; Other: Hydrolyzed whey protein; Other: Casein native; Other: Hydrolyzed casein; Other: Total milk protein native; Other: Hydrolyzed milk protein
- Hydrolyzed whey protein (Experimental): Hydrolyzed whey protein versus the 6 other arms
  Interventions: Other: Whey protein native; Other: Whey protein microgels; Other: Casein native; Other: Hydrolyzed casein; Other: Total milk protein native; Other: Hydrolyzed milk protein
- Casein native (Experimental): Casein native versus the 6 other arms
  Interventions: Other: Whey protein native; Other: Whey protein microgels; Other: Hydrolyzed whey protein; Other: Hydrolyzed casein; Other: Total milk protein native; Other: Hydrolyzed milk protein
- Hydrolyzed casein (Experimental): Hydrolyzed casein versus the 6 other arms
  Interventions: Other: Whey protein native; Other: Whey protein microgels; Other: Hydrolyzed whey protein; Other: Casein native; Other: Total milk protein native; Other: Hydrolyzed milk protein
- Total milk protein native (Experimental): Total milk protein native versus the 6 other arms
  Interventions: Other: Whey protein native; Other: Whey protein microgels; Other: Hydrolyzed whey protein; Other: Casein native; Other: Hydrolyzed casein; Other: Hydrolyzed milk protein
- Hydrolyzed milk protein (Experimental): Hydrolyzed milk protein versus the 6 other arms
  Interventions: Other: Whey protein native; Other: Whey protein microgels; Other: Hydrolyzed whey protein; Other: Casein native; Other: Hydrolyzed casein; Other: Total milk protein native

INTERVENTIONS:
Other: Whey protein native — Whey protein native against the 6 other arms
  Arms: Casein native; Hydrolyzed casein; Hydrolyzed milk protein; Hydrolyzed whey protein; Total milk protein native; Whey protein microgels
Other: Whey protein microgels — Whey protein microgels versus the six other arms
  Arms: Casein native; Hydrolyzed casein; Hydrolyzed milk protein; Hydrolyzed whey protein; Total milk protein native; Whey protein native
Other: Hydrolyzed whey protein — versus the six other arms
  Arms: Casein native; Hydrolyzed casein; Hydrolyzed milk protein; Total milk protein native; Whey protein microgels; Whey protein native
Other: Casein native — versus the six other arms
  Arms: Hydrolyzed casein; Hydrolyzed milk protein; Hydrolyzed whey protein; Total milk protein native; Whey protein microgels; Whey protein native
Other: Hydrolyzed casein — versus the six other arms
  Arms: Casein native; Hydrolyzed milk protein; Hydrolyzed whey protein; Total milk protein native; Whey protein microgels; Whey protein native
Other: Total milk protein native — versus the six other arms
  Arms: Casein native; Hydrolyzed casein; Hydrolyzed milk protein; Hydrolyzed whey protein; Whey protein microgels; Whey protein native
Other: Hydrolyzed milk protein — versus the six other arms
  Arms: Casein native; Hydrolyzed casein; Hydrolyzed whey protein; Total milk protein native; Whey protein microgels; Whey protein native

SUMMARY:
The purpose of the clinical study is to investigate the effect of the protein quality of high-protein meal replacements on the management of post-prandial blood glucose in healthy men.

DETAILED DESCRIPTION:
It was a double-blind, single center, randomized, crossover adaptive study design with 7 arms.

The subjects were submitted to 7 tests of ingestion of a high-protein meal replacement (test meal) in randomized order preferably a week apart. The 7 test meals were isocaloric, isonitrogenous and differed in their protein quality.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 50 years, male
* Healthy as determined by a medical questionnaire
* Normal weight: BMI 20 - 24.9 kg.m-2
* Normal fasting glycemia and insulinemia
* Normal fasting lipidemia (cholesterol and triglycerides)
* Normal liver function (transaminases, γ-GT) and kidney function (urea, creatinine)
* Capable of fast ingestion of the meal replacement (5-10 min)
* Having signed informed consent

Exclusion Criteria:

* Intestinal or metabolic diseases/disorders such as diabetic, renal, dyslipidemia, hepatic, hypertension, pancreatic or ulcer, including lacto-intolerance.
* Hypertension >150/95 mmHg
* Have had a gastrointestinal surgery
* Have a regular consumption of medication
* Vegetarian, vegan, under dietary supplements
* Have an alcohol intake: > 2 units a day or smoker
* Currently participating or having participated in a clinical trial during the last month
* Having given blood in the last month
* More than 5 x 45 min of intense exercise per week
* Volunteer who cannot be expected to comply with treatment

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Pouteau, Ph.D., Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- Nestec Clinical Development Unit / Metabolic Unit, Lausanne, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited among the Nestlé Research Center staff from June 2008 to May 2009
Pre-assignment Details: 25 healthy males were recruited; All presented all the inclusion criteria and none of the exclusion criteria listed in the protocol. The day before each test meal, the volunteers were recommended to eat normally as well as to conduct a normal physical activity. A standardized dinner was provided the night before testing.
Groups:
- 7 Proteins Were Tested Randomly: Seven high-protein meal replacement (MR) were tested. These high-protein MR contained 29% total energy intake (TEI) of protein, 28% TEI lipids and 43% TEI glucides in 400mL meal, were iso-nitrogenous and differed in their protein quality. The proteins were:
  * intact whey protein
  * whey protein micelles
  * exhaustively hydrolyzed whey protein
  * intact casein protein
  * exhaustively hydrolyzed casein protein
  * total milk protein
  * exhaustively hydrolyzed milk protein The high-protein MR were a 430g liquid meal containing 30g of the tested protein.
Period: 1st Protein Testing (1 Day)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 24 (1 subject withdrew his consent form before to starting the 1st intervention)
Completed | 24
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 24
Completed | 24
Not Completed | 0
Period: 2nd Protein Testing (1 Day)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 24
Completed | 24
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 24
Completed | 24
Not Completed | 0
Period: 3rd Protein Testing (1 Day)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 24
Completed | 24
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 24
Completed | 24
Not Completed | 0
Period: 4th Protein Testing (1 Day)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 24
Completed | 24
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: 5th Protein Testing (1 Day)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 23
Completed | 23
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 23
Completed | 23
Not Completed | 0
Period: 6th Protein Testing (1 Day)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 23
Completed | 23
Not Completed | 0
Period: Washout (7 Days)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 23
Completed | 23
Not Completed | 0
Period: 7th and Last Protein Testing (1 Day)
Arm/Group | 7 Proteins Were Tested Randomly
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants were recruited amoung the Nestlé Research Center staff.
Groups:
- Entire Study Population: Includes groups randomized to receive 7 products in a randomized series
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
Age Continuous [Mean (Standard Deviation); unit: Years] | 28.3 (1.5)
Age, Customized [Number; unit: participants]
  <=20 years | 0
  Between 20 and 50 years | 25
  >=50 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Region of Enrollment [Number; unit: participants]
  Switzerland | 25
Body weight [Mean (Standard Deviation); unit: kg] | 74.2 (1.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — BMI is obtained by dividing the weight (kg) by the square height (m2)
  kg/m2 | 23.5 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Post-prandial Plasma Responses of Glucose Concentrations
Description: The concentrations of glucose were analyzed in the 10 plasma samples collected over 3 h postprandially in all subjects (Baseline, 10, 20, 30, 45, 60, 90, 120, 150, and 180 min after product intake). The Area-Under-the-Curves (AUC) over 180 minutes from baseline were calculated by trapezoidal interpolation by excluding the area under baseline.
Time Frame: 180 minutes
Population: 23 subjects were investigated for AUC of glucose calculations
Measure: Mean (Standard Error); unit: mmole/L*min
Groups:
- Whey Protein Native; Whey Protein Microgels; Hydrolyzed Whey Protein; Casein Native; Hydrolyzed Casein; Total Milk Protein Native; Hydrolyzed Milk Protein: High-protein meal replacement : Acute ingestion of a high-protein meal replacement followed by blood sampling for 180 minutes.
Arm/Group | Whey Protein Native | Whey Protein Microgels | Hydrolyzed Whey Protein | Casein Native | Hydrolyzed Casein | Total Milk Protein Native | Hydrolyzed Milk Protein
Number analyzed (Participants) | 24 | 24 | 23 | 24 | 24 | 23 | 23
mmole/L*min | 136.5 (19) | 121.2 (13.1) | 102.9 (25.4) | 160.3 (18.6) | 88.7 (22.3) | 117.7 (15.6) | 121.5 (19.9)

2. Secondary Outcome: Post-prandial Plasma Responses of Glucagon, C-peptide, Amino Acids and Lipids
Time Frame: 180 minutes
Reporting Status: Not Posted

3. Primary Outcome: Calculation of the Area Under Curve Over Baseline for Plasma Insulin
Description: The concentrations of insulin were analyzed in the 10 plasma samples collected over 3 h postprandially in all subjects (Baseline, 10, 20, 30, 45, 60, 90, 120, 150, and 180 min after product intake). The Area-Under-the-Curves (AUC) over 180 minutes from baseline were calculated by trapezoidal interpolation by excluding the area under baseline.
Time Frame: 180 minutes from baseline
Measure: Mean (Standard Error); unit: nmole/L*min
Arm/Group | Whey Protein Native | Whey Protein Microgels | Hydrolyzed Whey Protein | Casein Native | Hydrolyzed Casein | Total Milk Protein Native | Hydrolyzed Milk Protein
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23 | 23
nmole/L*min | 34,428 (2,678) | 28,756 (2,383) | 32,319 (2,760) | 27,082 (2,283) | 34,847 (2,267) | 26,476 (1,699) | 37,922 (3,970)

ADVERSE EVENTS:
Arm/Group | Whey Protein Native | Whey Protein Microgels | Hydrolyzed Whey Protein | Casein Native | Hydrolyzed Casein | Total Milk Protein Native | Hydrolyzed Milk Protein
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/24 | 0/24 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/24 | 0/24 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No